CLINICAL TRIAL: NCT02743676
Title: Avian/Pandemic Influenza Registry
Brief Title: A Retrospective, Observational Registry of Participants With Avian Influenza Infection
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: NV22158
Record Dates: First submitted 2016-04-15; First posted 2016-04-19 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Influenza
Keywords: Avian Influenza
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Avian influenza A: Natural history of Avian influenza A, particularly H5N1 strain which has a high potential of causing a global human pandemic, and real-world treatment practices will be observed in this study. This registry program will not require, recommend, or provide any specific treatment or medications.

SUMMARY:
This is a global, multi-center, observational registry of participants with suspected or confirmed infection with avian influenza A H5N1. Data are collected through retrospective abstraction, from detailed case reports that may be published and available in the public domain, or as incident cases received directly from the treating physician or other medical personnel.

ELIGIBILITY:
Inclusion Criteria:

* Participants who develop influenza-like symptoms and who are considered to be epidemiologically linked by time, place, and exposure to a probable or confirmed avian influenza or human case of H5N1 infection are eligible for inclusion in the Registry. Cases with atypical symptom presentation (e.g., non-respiratory) are also included, in keeping with evolving knowledge about the clinical presentation of avian influenza.
* Participants with documented positive serological test who either remain asymptomatic or experience mild illness only
* Participants with laboratory confirmation of infection with influenza A (H5N1) who survive long enough to present for medical care

Exclusion Criteria:

- There are no exclusion criteria in this study

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective data are collected from participants with suspected or confirmed infection with avian influenza A H5N1.
Sampling Method: Probability Sample
Enrollment: 648 (Actual)
Dates: Start 2007-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with clinical outcome (death, recovery, or other overall clinical status) at the time of discharge from care | Up to 5 years

SECONDARY OUTCOMES:
Number of Participants with at least One Adverse Event (AE) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche